CLINICAL TRIAL: NCT02078232
Title: Randomized, Comparative Study of 19G Flex Versus 22G Standard Needles for Pancreatic Solid Tumors Diagnosis.
Brief Title: Comparison of Two Needles (19G Flex Versus 22G Standard) for Pancreatic Solid Tumors Diagnosis
Acronym: EASYFLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Society of Digestive Endoscopy (Other)
Responsible Party: Principal Investigator, Christian BOUSTIERE, MD, Head of Endoscopy Department, Hôpital Saint Joseph, Marseille, French Society of Digestive Endoscopy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SFED N°98
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-11

CONDITIONS: Adenocarcinoma of Head of Pancreas
Keywords: fine needle aspiration under ultrasound endoscopy; solid pancreatic tumors; head of pancreas; 19G Flex needle; 22G standard needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 19G flex needle puncture (Experimental): puncture of head of pancreas
  Interventions: Device: puncture of head of pancreas
- 22G needle puncture (Active Comparator): puncture of head of pancreas
  Interventions: Device: puncture of head of pancreas

INTERVENTIONS:
Device: puncture of head of pancreas — puncture of head of pancreatic solid mass with fine needle aspiration under endoscopic ultrasonographic control.
  randomization: puncture with either 22G needle or 19G flex needle
  Arms: 19G flex needle puncture
Device: puncture of head of pancreas — puncture of head of pancreatic solid mass with fine needle aspiration under endoscopic ultrasonographic control.
  randomization: puncture with either 22G needle or 19G flex needle
  Arms: 22G needle puncture

SUMMARY:
The purpose of this study is to compare the diagnostic gain between 22G standard needle vs 19G Flex needles transduodenal punctures of masses of the pancreatic head.

DETAILED DESCRIPTION:
The negative predictive value of fine needle aspiration under ultrasound endoscopy (EUS-FNA) for the diagnosis of solid pancreatic masses is about 70 - 80 % with the 22G standard needle. Pancreatic adenocarcinoma is known to have a severe prognosis and a low rate of survival even after curative surgery. The study of pancreatic solid tumors is one the main diagnostic problem present in the investigators daily practice. In most of non operated patients, EUS-FNA is the sole possibility to confirm the diagnosis of malignancy which is required to initiate chemotherapy and/or radiotherapy. To improve the performances of the EUS-FNA, new needles are now disposable either with a cutting window design (EchoTip ProCore-COOK Medical) or flexible 19G needle (19G Expect Flex - Boston-Scientific). The goal is to obtain more tissue material with the possibility of a histologic study without increasing the risk of the puncture which is very low (complications rate < 1%). The problem concerns the lesion of the head of the pancreas requiring a trans-duodenal access for the puncture . In this position, the needle is very difficult to push out the operator channel and, in some cases, the puncture is quite impossible with stiff needles as "ProCore" or standard 19G. Thus, the interest of flexible 19G needle is to be used in difficult technical cases as transduodenal access for head pancreatic tumors, with a good safety and more efficacy than 22G needles.

ELIGIBILITY:
Inclusion Criteria:

* patient with solid tumor of pancreas who has to receive a biopsy under endoscopic ultrasound (EUS)
* patient who understands the study procedures, risks and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria:

* patient who participates in an other study
* patient mentally or legally incapacitated
* patient with contraindications to the achievement of upper gastrointestinal endoscopy
* patient with haemorrhagic disease, disorder of hemostasis and coagulation (TP<60%, TCA>40sec and platelets <60000/mm3)
* patient with anticoagulant or antiaggregating treatment that could not be stopped for the endoscopic procedure
* patient with pancreatic cystic mass (fluid quota valued at more than 50% of the mass lesion on imaging)
* patient pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07-06 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
accuracy of 19G Flex Expect needle in the histological diagnosis of pancreatic solid tumors of the head of pancreas | 10 days
  accuracy and diagnostic gain of fine needle aspiration under ultrasound endoscopy (EUS-FNA) for the diagnosis of solid pancreatic tumors of the head of pancreas: comparison between 19G Flex and 22G standard needles punctures.

SECONDARY OUTCOMES:
morbidity | 2 minutes, up to day 30
  immediate per-procedure complications and delayed morbidity (up to day 30) side effects resulting of technical failure or dysfunction of the puncture ease of handling for the two needles (visual analogic scale)
quality of histology | 10 days
  quality of histological specimens obtained with the 2 types of needles (visual analogic scale)

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTIAN BOUSTIERE, MD, Principal Investigator — FRENCH SDE
Locations (1):
- Hopital Saint Joseph, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenssen C, Dietrich CF. Endoscopic ultrasound-guided fine-needle aspiration biopsy and trucut biopsy in gastroenterology - An overview. Best Pract Res Clin Gastroenterol. 2009;23(5):743-59. doi: 10.1016/j.bpg.2009.05.006. PMID 19744637
- [Background] Takemoto T, Aibe T, Fuji T, Okita K. Endoscopic ultrasonography. Clin Gastroenterol. 1986 Apr;15(2):305-19. PMID 3524913
- [Background] Erickson RA. EUS-guided FNA. Gastrointest Endosc. 2004 Aug;60(2):267-79. doi: 10.1016/s0016-5107(04)01529-9. No abstract available. PMID 15278063
- [Background] Hewitt MJ, McPhail MJ, Possamai L, Dhar A, Vlavianos P, Monahan KJ. EUS-guided FNA for diagnosis of solid pancreatic neoplasms: a meta-analysis. Gastrointest Endosc. 2012 Feb;75(2):319-31. doi: 10.1016/j.gie.2011.08.049. PMID 22248600
- [Background] Song TJ, Kim JH, Lee SS, Eum JB, Moon SH, Park DY, Seo DW, Lee SK, Jang SJ, Yun SC, Kim MH. The prospective randomized, controlled trial of endoscopic ultrasound-guided fine-needle aspiration using 22G and 19G aspiration needles for solid pancreatic or peripancreatic masses. Am J Gastroenterol. 2010 Aug;105(8):1739-45. doi: 10.1038/ajg.2010.108. Epub 2010 Mar 9. PMID 20216532
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Adler DG, Jacobson BC, Davila RE, Hirota WK, Leighton JA, Qureshi WA, Rajan E, Zuckerman MJ, Fanelli RD, Baron TH, Faigel DO; ASGE. ASGE guideline: complications of EUS. Gastrointest Endosc. 2005 Jan;61(1):8-12. doi: 10.1016/s0016-5107(04)02393-4. PMID 15672049
- [Background] Al-Haddad M, Wallace MB, Woodward TA, Gross SA, Hodgens CM, Toton RD, Raimondo M. The safety of fine-needle aspiration guided by endoscopic ultrasound: a prospective study. Endoscopy. 2008 Mar;40(3):204-8. doi: 10.1055/s-2007-995336. Epub 2007 Dec 4. PMID 18058615
- [Background] Carrara S, Arcidiacono PG, Mezzi G, Petrone MC, Boemo C, Testoni PA. Pancreatic endoscopic ultrasound-guided fine needle aspiration: complication rate and clinical course in a single centre. Dig Liver Dis. 2010 Jul;42(7):520-3. doi: 10.1016/j.dld.2009.10.002. Epub 2009 Dec 1. PMID 19955025
- [Background] Boustiere C, Veitch A, Vanbiervliet G, Bulois P, Deprez P, Laquiere A, Laugier R, Lesur G, Mosler P, Nalet B, Napoleon B, Rembacken B, Ajzenberg N, Collet JP, Baron T, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Endoscopy and antiplatelet agents. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2011 May;43(5):445-61. doi: 10.1055/s-0030-1256317. Epub 2011 May 4. PMID 21547880
- [Background] Fayers PM, Machin D. Sample size: how many patients are necessary? Br J Cancer. 1995 Jul;72(1):1-9. doi: 10.1038/bjc.1995.268. PMID 7599035
- [Derived] Laquiere A, Lefort C, Maire F, Aubert A, Gincul R, Prat F, Grandval P, Croizet O, Boulant J, Vanbiervliet G, Penaranda G, Lecomte L, Napoleon B, Boustiere C. 19 G nitinol needle versus 22 G needle for transduodenal endoscopic ultrasound-guided sampling of pancreatic solid masses: a randomized study. Endoscopy. 2019 May;51(5):436-443. doi: 10.1055/a-0757-7714. Epub 2018 Nov 19. PMID 30453379